CLINICAL TRIAL: NCT07341906
Title: Evaluation of the Contribution of Artificiel Inteligence on a Dermatologist Tele -Expertise Request Made by General Praticioner : a Retrospective and Single-center Study.
Brief Title: Diagnosis Evaluation Made by Artificial Inteligence in Response to a Request Made by General Praticioner on OMNIDOC to the Dermatologist of the CHU of Nice. A Comparison of This Response by the One Made by the Dermatologist.
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25MedInterne01
Record Dates: First submitted 2025-12-24; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Skin Diseases; Artificial Intelligence
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Expert opinion: The expert had provided a diagnosis and a support based on the guideline in France
  Interventions: Other: The diagnosis made by Chat Gpt
- chatGPT opinion: ChatGPT will provide a diagnosis and the support based on the guideline in France
  Interventions: Other: The diagnosis made by Chat Gpt
- Specialized AI opinion: Specialised IA will provide a diagnosis and the support based on the guideline in France
  Interventions: Other: The diagnosis made by Chat Gpt

INTERVENTIONS:
Other: The diagnosis made by Chat Gpt — The expert had provided a diagnosis and a support based on the guideline in France

SUMMARY:
The First part of the study will be the inclusion of our patients (those for whom a tele-expertise request has been made by their general practitioner on the OMNIDOC platform between the 1st of May 2024 and the 31st of December 2025. ) After that, the team will investigate the non opposition patient to the use of their personal information.

Subsequently, the clinical study will focus on comparing the diagnosis made by chat gpt expert and a dermatologist from the University Hospital of Nice to a request of dermatology tele-expertise made by general praticioner on OMNIDOC

ELIGIBILITY:
Inclusion Criteria:

* Adult with a request on OMNIDOC made by their general practitioner.
* Adult not opposed Social Security affiliation.
* Diagnosis made by a dermatologist.

Exclusion Criteria:

* Pediatric case.
* Unusable image.
* Absence of diagnosis made by a dermatologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient for whom a tele-expertise request has ben made by their general practitioner on the OMNIDOC platform between the 1st of May 2024 and the 31st of December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare the diagnoses offered by artificial intelligence to those proposed by the experts on requests for tele-expertise. | From 01 May 2025 - 31 December 2026
  Check the correspondence between the diagnosis made by the expert and the artificial intelligence on the photos, the diagnosis and supports.

SECONDARY OUTCOMES:
Compare the support and response times offered by artificial intelligence to those offered by experts for dermatology tele-expertise requests. | From 01 May 2025 - 31 December 2026
  Check the consistency between the expert's instructions and the timeframe for intervention, and the information provided by the two artifical intelligence by The photos, the diagnosis and supports
Compare the differences between the responses offered by chatGPT and the specific dermatologic artificial intelligence | From 01 May 2025 - 31 December 2026
  Compare the differences between the responses offered by chatGPT and the specific dermatologic artificial intelligence by the photos, the diagnosis and supports

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Alpes Maritimes, France